CLINICAL TRIAL: NCT03052010
Title: Delivery of Integrated PrEP and ART for Couples in Kenya
Brief Title: The Partners Scale-Up Project
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); Kenya National AIDS & STI Control Programme (Other); National Institute of Mental Health (NIMH) (NIH); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Jared Baeten, Professor, Global Health, Medicine, & Epidemiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002183; 2R01MH095507 (NIH)
Record Dates: First submitted 2017-02-05; First posted 2017-02-14 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: HIV-1-infection
Keywords: HIV-1 serodiscordant couples; PrEP as Bridge to ART

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP for HIV-1 uninfected partners and ART for HIV-1 infected (Other): Integrated PrEP as a bridge to ART HIV-1 prevention strategy
  Interventions: Other: Integrated PrEP as a bridge to ART HIV-1 prevention strategy; Drug: PrEP; Drug: ART

INTERVENTIONS:
Other: Integrated PrEP as a bridge to ART HIV-1 prevention strategy — The PrEP as a bridge to ART intervention will be introduced into clinics according to Kenya national guidelines using a stepped wedge design, stratified by region. The components of the intervention are: a) Couples' HIV-1 counseling and testing; 2) PrEP as a bridge to ART: PrEP offered prior to ART initiation in couples in which the HIV-1 infected partner is not on ART due to refusal/delay, during the first 6 months after ART start during viral decline, and then discontinuation; 3) ART at any CD4 count, offered to all HIV-1 infected partners, with ongoing promotion/counseling for those delaying/declining;4) Standard of care HIV-1 prevention services
Drug: PrEP — A fixed-dose, oral co-formulation of emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) is the approved and preferred regimen for HIV-1 prevention in Kenya and the United States. The World Health Organization (WHO) recommends TDF-containing medications as PrEP, which includes TDF combined with FTC as well as potentially TDF alone and TDF combined with lamivudine (or 3TC, a medication closely related to FTC). Any TDF-containing medications that align with WHO and Kenya national guidelines for PrEP will be used. PrEP medication will come from clinic stocks.
Drug: ART — ART medications will be provided according to Kenya national ART policies and will come from clinic stocks.

SUMMARY:
An implementation project to scale-up delivery of antiretroviral-based HIV-1 prevention methods to Kenyan HIV-1 serodiscordant couples in HIV-1 care centers. Pre-exposure prophylaxis (PrEP) as a bridge to antiretroviral therapy (ART) HIV-1 prevention strategy will be introduced into 24 public HIV-1 care centers in central and western Kenya according to national guidelines using a stepped wedge design, stratified by region.

DETAILED DESCRIPTION:
PrEP as a bridge to ART strategy will be introduced into 24 Kenyan public HIV-1 care centers according to national guidelines, in staged fashion, stratified by region (a stepped wedge design). Monitoring and evaluation activities will identify implementation barriers and solutions, characterize costs, and provide best practices for further scale-up. A research component will establish prospective open cohorts of couples at each clinic (up to 200) to study how the program is effectively implemented. Follow-up in the cohorts will be for up to 36 months at each care center and will evaluate impact, costs, and facilitators and barriers to implementation at patient, provider and health system levels.

ELIGIBILITY:
Inclusion Criteria:

* For HIV-1 uninfected members of the couple
* Age ≥18
* Able and willing to provide consent for follow-up in the cohort
* HIV-1 uninfected based on negative HIV-1 tests, per Kenya national guidelines
* Not currently using PrEP

For HIV-1 infected members of the couple

* Age ≥18
* Able and willing to provide consent for follow-up in the cohort
* HIV-1 infected based on positive HIV-1 tests, per Kenya national guidelines
* Not currently using ART

For both members of the couple - Meet criteria for initiating PrEP as per Kenya national guidelines, including:

* HIV-1 infected member not currently using ART, on ART <6 months, or on ART but not virally suppressed based on a viral load test done at the clinic as per Kenya national guidelines or
* Trying to conceive

For key delivery informants

- Able and willing to provide consent

Exclusion Criteria:

* Otherwise not eligible based on the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4898 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of HIV-1 infected persons whose partners are tested for HIV-1 before/after PrEP as a bridge to ART is implemented | up to 36 months
PrEP initiation | up to 36 months
  Measure the number of HIV-1 uninfected partners initiating PrEP.
PrEP adherence | up to 6 months
  Adherence by HIV-1 uninfected partners until their HIV-1 infected partners initiate ART and sustain use for six months. Adherence will be measured by self reported and random dry blood spot for tenofovir levels
HIV-1 uninfected partners staying HIV-1 uninfected. | up to 36 months
ART initiation | up to 36 months
  Number of HIV-1 infected partners newly initiating ART
ART adherence | up to 6 months
  Adherence measured by plasma RNA viral load. Viral load will be abstract from the HIV-infected partners records.
Facilitators and barriers to implementation of integrated PrEP and ART | up to 36 months
  Mixed methods assessment of how integrated PrEP and ART is implemented at the level of provider, health center, and health systems
PrEP delivery operational tools | 24 months
  Training manual on deliver of integrated PrEP and ART HIV prevention strategy for couples will be developed.
Cost and cost-effectiveness of the integrated PrEP and ART when delivered in public health clinics. | up to 36 months
  Time and motions to define the cost and cost-effectiveness of intervention summarized in terms of HIV infections averted, disability-adjusted life years saved, and incremental cost-effectiveness over routine HIV-1 care

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baeten, MD, PhD, Principal Investigator — University of Washington; Kenneth K. Mugwanya, MBChB, MS, PhD, Study Director — University of Washington
Locations (2):
- Kenya (2):
  - KEMRI, Kisumu
  - Partners in Health Research and Development, Thika

IPD SHARING:
Plan to Share IPD: Yes
Data from the Partners Scale-Up Project will be available at end of the Project by contacting the International Clinical Research Center at the University of Washington (icrc@uw.edu)

REFERENCES:
- [Derived] Irungu EM, Mugwanya KK, Mugo NR, Bukusi EA, Donnell D, Odoyo J, Wamoni E, Peacock S, Morton JF, Ngure K, Mugambi M, Mukui I, O'Malley G, Baeten JM; Partners Scale-Up Project Team. Integration of pre-exposure prophylaxis services into public HIV care clinics in Kenya: a pragmatic stepped-wedge randomised trial. Lancet Glob Health. 2021 Dec;9(12):e1730-e1739. doi: 10.1016/S2214-109X(21)00391-0. PMID 34798031
- [Derived] Irungu EM, Odoyo J, Wamoni E, Bukusi EA, Mugo NR, Ngure K, Morton JF, Mugwanya KK, Baeten JM, O'Malley G; Partners Scale-Up Project Team. Process evaluation of PrEP implementation in Kenya: adaptation of practices and contextual modifications in public HIV care clinics. J Int AIDS Soc. 2021 Sep;24(9):e25799. doi: 10.1002/jia2.25799. PMID 34496148
- [Derived] Peebles K, Mugwanya KK, Irungu E, Odoyo J, Wamoni E, Morton JF, Ngure K, Bukusi EA, Mugo NR, Masyuko S, Mukui I, Baeten JM, Barnabas RV; Partners Scale-Up Project Team. Low costs and opportunities for efficiency: a cost analysis of the first year of programmatic PrEP delivery in Kenya's public sector. BMC Health Serv Res. 2021 Aug 16;21(1):823. doi: 10.1186/s12913-021-06832-3. PMID 34399736
- [Derived] Irungu EM, Ngure K, Mugwanya K, Mugo N, Bukusi E, Wamoni E, Odoyo J, Morton JF, Bernabee G, Mambo B, Masyuko S, Mukui I, O'Malley G, Baeten JM. Training health care providers to provide PrEP for HIV serodiscordant couples attending public health facilities in Kenya. Glob Public Health. 2019 Oct;14(10):1524-1534. doi: 10.1080/17441692.2019.1588908. Epub 2019 Mar 14. PMID 30871413
- [Derived] Mugwanya KK, Irungu E, Bukusi E, Mugo NR, Odoyo J, Wamoni E, Ngure K, Morton JF, Peebles K, Masyuko S, Barnabee G, Donnell D, Barnabas R, Haberer J, O'Malley G, Baeten JM; Partners Scale Up Team. Scale up of PrEP integrated in public health HIV care clinics: a protocol for a stepped-wedge cluster-randomized rollout in Kenya. Implement Sci. 2018 Sep 4;13(1):118. doi: 10.1186/s13012-018-0809-7. PMID 30180860